CLINICAL TRIAL: NCT00003357
Title: Vaccination of High Risk Breast Cancer Patients Lacking Identifiable Disease With GM2-KLH Conjugate Plus the Immunological Adjuvant QS21
Brief Title: Vaccine Therapy Plus QS21 in Treating Women With Breast Cancer Who Have No Evidence of Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-123; MSKCC-97123; NCI-H98-0015
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — saponin QA-21V1

INTERVENTIONS:
Biological: GM2-KLH vaccine
Biological: QS21

SUMMARY:
RATIONALE: Vaccines made from GM2-KLH and given with QS21 may make the body build an immune response to and kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of GM2-KLH vaccine plus QS21 in treating patients with breast cancer who have no evidence of disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether immunization with GM2-KLH vaccine plus the immunological adjuvant QS21 induces an antibody response against GM2 and cells expressing GM2 in disease free patients at high risk for recurrence of breast cancer.

OUTLINE: GM2-KLH vaccine plus QS21 is administered subcutaneously to sites on the upper arm and upper leg at weekly intervals for 4 weeks. Two additional vaccines are administered at weeks 12 and 24. Patients are followed every 3 months after the sixth vaccination.

PROJECTED ACCRUAL: A total of 9 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Eligible patients must have no evidence of disease in addition to 1 of the following features: Stage I, II, or III breast cancer and have received adjuvant chemotherapy and remain clinically free of identifiable disease, but have rising CA15.3 (BR2729) or CEA levels Stage III breast cancer and have completed adjuvant therapy no more than 24 months ago Recurrence in the ipsilateral axilla following a lumpectomy/axillary dissection or modified radical mastectomy Recurrence in the ipsilateral breast following a lumpectomy/axillary dissection Stage II breast cancer with at least 4 positive axillary lymph nodes at 24 months following completion of adjuvant therapy Patients with isolated elevation of the CEA level must have a colonoscopy to rule out colon carcinoma A colonoscopy within the past 5 years is acceptable if there is no strong family history of colon carcinoma, colonic polyps, or inflammatory bowel disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Premenopausal or postmenopausal Performance status: Karnofsky 90-100% Life expectancy: Not specified Hematopoietic: Lymphocyte count at least 500/mm3 WBC count at least 3,000/mm3 Hepatic: Aspartate aminotransferase no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No New York Heart Association class III or IV cardiac disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other concurrent active cancers except basal cell or squamous cell carcinomas of the skin No history of a seafood allergy No known history of immunodeficiency or autoimmune disease

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: No concurrent steroids Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 4 weeks since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 1998-01; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Ann Gilewski, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States